CLINICAL TRIAL: NCT07349381
Title: An Open-label, Randomized, Multiple-dose, Two-cycle, Two-way Crossover Phase 1 Study to Evaluate the Effect of Food on the Pharmacokinetics of CX11 Tablets in Healthy Participants
Brief Title: A Food-Effect Study of CX11 in Healthy Participants
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Vincentage Pharma Co., Ltd (Industry)
Collaborators: Corxel Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CX11101
Record Dates: First submitted 2026-01-08; First posted 2026-01-16 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Obesity & Overweight; Type 2 Diabetes
MeSH Terms: conditions — Obesity; Overweight; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Fasted-Fed Arm (Experimental): Fasted-Fed Group
  Interventions: Drug: CX11 (VCT220)
- Fed-Fasted Arm (Experimental): Fed-Fasted Group
  Interventions: Drug: CX11 (VCT220)

INTERVENTIONS:
Drug: CX11 (VCT220) — CX11 (VCT220) administered orally to participants who are in fasted/fed state in the first 6 consecutive days, and in fed/fasted state on the 7th day

SUMMARY:
This study is to evaluate the food effect (FE) on the PK of 200 mg CX11 in healthy participants

ELIGIBILITY:
Inclusion Criteria:

1. Fully understand the objective, nature, methods, and possible adverse reactions of the study; be able to communicate well with the investigator; voluntarily take part in the study and be willing to comply with the requirements of this study; and sign the informed consent form before all study procedures are started
2. Weight ≥ 50.0 kg for men and ≥ 45.0 kg for women, and body mass index (BMI) is ≥ 20.0 kg/m2 and < 28 kg/m2 at the screening visit and on Day 21.

Exclusion Criteria:

1. Participants with allergic constitution or known previous history of allergy to CX11 or similar compounds and related excipients, or history of atopic allergic diseases
2. Participants who have experienced clinically significant acute diseases during the pre-study screening period or within 2 weeks prior to the first dose of the investigational product
3. Participants who have pre-existing condition interfering with normal gastrointestinal anatomy or motility, hepatic and/or renal function that could affect drug absorption, distribution, metabolism, and/or excretion as judged by the investigator, or plan to receive any surgery during the study
4. Participants suffering from any clinically significant chronic diseases, including but not limited to disorders of the respiratory system, cardiovascular system, urinary system, blood system, endocrine system, and immune system, as well as the digestive system (e.g., history of or current fatty liver disease, including metabolic dysfunction-associated steatohepatitis
5. History of thyroid dysfunction requiring medication or with a thyroid stimulating hormone (TSH) level exceeding the normal reference range at screening or on Day 21
6. Participants who have been vaccinated within 30 days before the screening or plan to be vaccinated during the study
7. Participated in any other clinical study and received an investigational intervention within 90 days or 5 elimination half-lives (whichever is longer) of the investigational intervention, prior to screening

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2026-03-26 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Area Under the Concentration-time curve from 0 to 24 hour (AUC0-24) of CX11 (VCT220) | Predose at Day1 up to 35 days postdose
  AUC0-24 of of CX11 (VCT220)
Maximum Observed Concentration (Cmax) of CX11 (VCT220) | Predose at Day1 up to 35 days postdose
  Cmax of CX11 (VCT220)
Time to Maximum Observed Concentration (Tmax) of CX11 (VCT220) | Predose at Day 1 up to 35 days postdose
  Tmax of CX11 (VCT220)

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Xuhui Central Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No